CLINICAL TRIAL: NCT01602250
Title: Prevention of Systemic Toxicity Induced by Levobupivacaine and Ropivacaine by Intralipid®
Brief Title: Local Anaesthetics Toxicity and Intralipid®
Acronym: TOXALIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P100501
Record Dates: First submitted 2012-02-23; First posted 2012-05-18 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Toxicity; Adverse Effects
Keywords: Anesthetics, local; Toxicity; Adverse effects
MeSH Terms: interventions — Levobupivacaine; Ropivacaine; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- levobupivacaine placebo (Placebo Comparator): levobupivacaine placebo
  Interventions: Drug: placebo
- levobupivacaine Intralipid® (Experimental): levobupivacaine Intralipid®
  Interventions: Drug: Intralipid®
- ropivacaine Intralipid® (Experimental): ropivacaine Intralipid®
  Interventions: Drug: Intralipid®
- ropivacaine placebo (Placebo Comparator): ropivacaine placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Levobupivacaine 8 mg/min ropivacaine 8 mg/min
  Other Names: levobupivacaine; ropivacaine
  Arms: levobupivacaine placebo; ropivacaine placebo
Drug: Intralipid® — Levobupivacaine 8 mg/min ropivacaine 8 mg/min Intralipid® 120 ml in one min
  Arms: levobupivacaine Intralipid®; ropivacaine Intralipid®

SUMMARY:
The systemic toxicity of local anaesthetics may be treated using lipid emulsions ("lipid rescue"). However, there is no evidence-based proof of the efficacy of the treatment. The aim of the intended protocol is to study the effect of the emulsion Intralipid® on the toxicity prodromes in volunteers receiving either levobupivacaine or ropivacaine. After a sensitization session with lidocaine, subjects will receive in a double blind, crossover manner an i.v. infusion of levobupivacaine or ropivacaine followed by a rapid infusion of Intralipid®. The primary outcome will be the time of appearance of early neurologic signs of toxicity. In addition, the EEG and ECG will be monitored and blood sampling will be performed in order to evaluate the changes in pharmacokinetics induced by the emulsion.

DETAILED DESCRIPTION:
Regional anaesthesia may induce toxic neurologic and cardiac reactions related to inadvertent intravenous injection or rapid absorption of local anaesthetics. Despite the appearance of the less toxic agents ropivacaine and levobupivacaine, the problem remains. Recently, a new therapeutics called "lipid rescue" emerged. This rapid injection of a lipid emulsion is supposed to act as a lipid sink, thus delaying the release of the toxic molecules to the target organs. Animal studies as well as clinical reports seem to favour this treatment. However, there is no evidence-based proof of the efficacy of this "lipid rescue".

The aim of the study is 1) to verify the efficacy of a lipid emulsion (Intralipid® 20%) on the toxicity induced by the local anaesthetics ropivacaine and levobupivacaine and 2) to compare the effect of the emulsion on the two agents.

Sixteen volunteers with strictly normal ECG and EEG will participate to the study.

After a sensitization session with lidocaine, the subjects will receive levobupivacaine or ropivacaine i.v. at a rate of 8 mg/min (max 120 mg) followed two minutes after the beginning of infusion by a bolus injection of Intralipid® 20% or of saline 120 mL in 1 minute. The infusion of local anaesthetics will be stopped immediately at the appearance of the early signs of toxicity. In addition to the recognition of the signs by the subject (trained by the sensitization session), an anaesthesiologist will ask if the subject has any symptom. A continuous monitoring of the EEG and of the ECG will be performed.

Sixteen subjects completing the study have been considered necessary to achieve a power of 90 % with an alpha risk of 5 %. A mean time to first signs of 3.8 ± 1.2 min has been considered in the placebo groups. A 45 % difference in the primary outcome has been considered. The study will be double blind crossover as a Latin square (four treatments, four sessions, four replications).

The investigators will consider the time between infusion initiation and appearance of the early signs of toxicity as primary outcome. The secondary outcomes will be the changes in ECG and EEG variables and the pharmacokinetic parameters observed. For that purpose, blood will be sampled until the 8th hour after the beginning of local anaesthetic infusion.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers ASA1

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Duration of drug infusion | less than 15 minutes

SECONDARY OUTCOMES:
EEG : electroencephalogram | < 15 minutes
  Detection of sub-clinical seizure activity
ECG : electrocardiogram | < 15 minutes
  Duration of PR, QRs intervals
pharmacokinetics of local anesthetics (Area under the plasma concentration versus time curve (AUC)) | 8 h
  blood concentration of local anesthetics during 8 hours post administration : Area under the plasma concentration versus time curve (AUC)"

CONTACTS AND LOCATIONS:
Overall Officials: Dan Benhamou, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CIC plurithématique Paris-Est (CIC-9304), Paris, France

REFERENCES:
- [Result] Dureau P, Charbit B, Nicolas N, Benhamou D, Mazoit JX. Effect of Intralipid(R) on the Dose of Ropivacaine or Levobupivacaine Tolerated by Volunteers: A Clinical and Pharmacokinetic Study. Anesthesiology. 2016 Sep;125(3):474-83. doi: 10.1097/ALN.0000000000001230. PMID 27404223